CLINICAL TRIAL: NCT05826613
Title: Respiratory Registry for Lung Health: a Prospective, Observational Study on Adult Patients With Asthma or COPD for the Identification of Genetic Biomarkers Related to the Chronic Obstructive Lung Diseases
Brief Title: Respiratory Registry for Lung Health: a Prospective, Observational Study on Adult Patients With Asthma or COPD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Responsible Party: Sponsor
Other Study IDs: ESR-18-13818
Record Dates: First submitted 2023-03-14; First posted 2023-04-24 (Actual); Last update posted 2023-04-24 (Actual); Status verified 2023-03

CONDITIONS: Chronic Obstructive Pulmonary Disease; Asthma
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Asthma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples With DNA — Blood, serum, sputum, urine, stool, lung biopsies, bronchoaspirate and bronchoalveolar lavage specimens
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- adults with COPD and asthma: Male or female aged >18 years with clinical diagnosis of either COPD or asthma.

SUMMARY:
The database will contain a wide range of demographic, clinical, radiological, laboratory, functional, microbiological, treatment, and clinical outcomes data on adults with chronic obstructive pulmonary disease (COPD) and asthma enrolled during stable state with annual follow-up (either one or two-year follow up).

Primary Objective: To collect clinical (including quality of life measurements), laboratory (including non-invasive measurement of biomarkers), microbiological, radiological, functional, treatment variables and clinical outcomes, in adult patients with either asthma or COPD during stable state.

Secondary Objectives: To identify genetic and other omics patterns to develop phenotype handprints for adults with either asthma or COPD. To characterize the airways microbiome in stable patients with either asthma or COPD and identify correlation with clinical phenotypes and/or endotypes.

DETAILED DESCRIPTION:
Currently, the World Health Organization estimates that chronic obstructive pulmonary disease (COPD) affects 65 million individuals worldwide and asthma affects 235 million. (World Health Organization. Chronic respiratory diseases. URL: http://www.who.int/respiratory/en/). In 2015, mortality from COPD exceeded 3 million deaths, while mortality from asthma included approximately 400 000 deaths (1). Unquestionably, COPD and asthma pose a significant global burden to which many of our healthcare resources are devoted.

COPD pathology is thought to be primarily due to inflammation. However, Eapen et al.(2) found a reduction in total cellularity in both large (endobronchial biopsies) and small airways (resected lung tissues) with a corresponding reduction in key innate inflammatory cell populations in mild-moderate COPD patients. Colonizing microbes were also found to contribute to pathogenesis, with a possible mechanism through perpetuation of negative immune responses over time (3).

Although cigarette smoking is the most significant risk factor, only a fraction of smokers develops COPD, so genetic associations should also be considered when assessing potential risk factors. The knowledge of the pathogenic mechanisms and genetic bases of respiratory diseases is fundamental for the correct setting of pharmacological and non-pharmacological management. If we consider the main respiratory diseases (COPD, asthma, idiopathic pulmonary fibrosis) but also the so-called rare diseases (e.g. cystic fibrosis), it is evident that both the expression of the disease and the response to treatment are very different among patients. Recent evidences have shown that these responses are related to different genetic models. Decision-making in medical care for decades has often relied on a "one-size-fits-all" approach that applies mean-effect-size results from studies to individual patients. The goal of precision medicine, in contrast, is to allow for more accurate treatment and prevention, decisions based on matching a patient's exposure, lifestyle and biological profile to that of similar patients with measured outcomes. It could be reasonable to hypothesize that mutations in genes which are involved in other respiratory diseases (such as primary ciliary dyskinesia or cystic fibrosis) might be present also in patients with either asthma or COPD. These mutations might alter the function of specific proteins (such as the cystic fibrosis transmembrane conductance regulator protein) and, thus, contribute to the pathophysiology of asthma or COPD. The goal of many "-omics" studies thus far has been to build a knowledgebase of omic variation using single-technology approaches that will help enable precision medicine by providing reference data to identify groups of individuals who share various attributes. In addition to collecting omics data, the application of sophisticated algorithms and use of extensive computational resources to integrate datasets are required to fully characterize diverse patients. The Respiratory Registry project aims to describe the epidemiology of chronic respiratory diseases, including COPD and Asthma, in the cities of Milan, Bergamo and Rome, to define different clinical phenotypes of these diseases, the relative genetic models and the endotypic expression, and then propose new therapeutic approaches, through the implementation of a clinical registry and an enlarged genetic study.

A database of respiratory diseases would have many important functions including but not limited to: 1) Analysis and evaluation of current standard operating procedures in different centres in Milan, Bergamo and Rome in order to compare them with recommendations of the international guidelines and with those used in other countries; 2) Analysis and assessment of differences in the management of adult patients by various professionals in the different centres in order to identify any area of improvement and/or the need to perform further clinical or translation studies; 3) Analysis and evaluation of several factors of disease severity (e.g., recurrence, hospitalization, mortality) that require large amounts of data not obtainable from monocentric studies.

The database will contain a wide range of demographic, clinical, radiological, laboratory, functional, microbiological, treatment, and clinical outcomes data on adults with COPD and asthma enrolled during stable state with annual follow-up (either one or two-year follow up). The database will be developed at the Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico di Milano and managed by the University Pneumology Unit of this hospital (Promoter of the study). Other University Pneumology Units will be involved, including those from the ASST Santi Paolo e Carlo Hospital in Milan, the ASST Fatebenefratelli-Sacco Hospital in Milan, the IRCCS Policlinico San Donato Hospital in San Donato, Milan, the Papa Giovanni XXIII Hospital in Bergamo and the Respiratory Unit of the Policlinico Gemelli in Rome. Data will be recorded using a case report form (CRF), incorporating all the variables related to the obstructive respiratory diseases identified as relevant for the purpose of this study: COPD and asthma. Study participants will also enter patient follow-up data on an annual basis to provide longitudinal data regarding clinical and therapeutic changes, as well as clinical outcomes. The total study duration will be 3 years, including 2 years for enrollment and at least 1 year of follow-up.

The study will be conducted in accordance with the principles of Good Clinical Practice (GCP). A favourable ethical opinion will be obtained first (as coordinating centre) by the Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico in Milan and then by each partner site from the appropriate research ethics committee. Furthermore, any other necessary approval required by partner site will be obtained prior to the commencement of the study at that site. All patients must provide written consent to participate in the registry. It is the responsibility of the investigator at each centre to obtain the appropriate local approvals. This prospective observational study will provide important data for the personalised management of obstructive lung diseases. No risk for the patient is foreseen. Informed consent for participation in the study, sample collection and omic analyses will be mandatory.

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent prior to any study specific procedures.
* Male or Female aged > 18 years.
* Clinical Diagnosis of either COPD or Asthma

Exclusion Criteria:

* No specific exclusion criteria will be applied to the registry in order to be as adherent as possible to the real-life population

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male or Female aged > 18 years with clinical Diagnosis of either COPD or Asthma.
  Asthma and COPD will be defined according to the latest international guidelines (https://goldcopd.org and https://ginasthma.org/2018-gina-report-global-strategy-for-asthmamanagement-and-prevention/)
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2019-09-10 (Actual); Primary Completion 2024-05-31 (Estimated); Study Completion 2024-05-31 (Estimated)

PRIMARY OUTCOMES:
Auscultation of the chest | 1 year
  A respiratory physical examination, according to the usual care, will be performed and include an assessment of the following: presence of wheeze (yes or no), presence of stridor (yes or no), presence of crackles (yes or no).
Presence of dyspnoea (mMRC scale) | 1 year
  A respiratory physical examination, according to the usual care, will be performed and include an assessment of the presence of dyspnoea. The measurement that will be used to assess this outcome measure is mMRC scale.
Forced vital capacity (FVC) | 1 year
  A complete respiratory functional evaluation will be performed according to the usual care for COPD and Asthma patient. Pulmonary function testing will include: FVC (reported in l)
Forced Expiratory Volume in the 1st second (FEV1) | 1 year
  A complete respiratory functional evaluation will be performed according to the usual care for COPD and Asthma patient. Pulmonary function testing will include: FEV1 (reported in l)
Peak expiratory flow (PEF) | 1 year
  A complete respiratory functional evaluation will be performed according to the usual care for COPD and Asthma patient. Pulmonary function testing will include: PEF(reported in l/min)
Vital capacity (VC) | 1 year
  A complete respiratory functional evaluation will be performed according to the usual care for COPD and Asthma patient. Pulmonary function testing will include: VC (reported in l)
Total Lung Capacity (TLC) | 1 year
  A complete respiratory functional evaluation will be performed according to the usual care for COPD and Asthma patient. Pulmonary function testing will include: TLC (reported in l)
Residual Volume (RV) | 1 year
  A complete respiratory functional evaluation will be performed according to the usual care for COPD and Asthma patient. Pulmonary function testing will include: RV (reported in l)
specific airway resistance (SRaw) | 1 year
  A complete respiratory functional evaluation will be performed according to the usual care for COPD and Asthma patient. Pulmonary function testing will include: sRaw (reported in kPa)
specific airway conductance (SGaw) | 1 year
  A complete respiratory functional evaluation will be performed according to the usual care for COPD and Asthma patient. Pulmonary function testing will include: sGaw (reported in kPa)
Diffusing Capacity Of The Lungs For Carbon Monoxide (DLCO) | 1 year
  A complete respiratory functional evaluation will be performed according to the usual care for COPD and Asthma patient. Pulmonary function testing will include: DLCO.
fraction of exhaled NO (FENO) | 1 year
  A complete respiratory functional evaluation will be performed according to the usual care for COPD and Asthma patient. Pulmonary function testing will include: FeNO.
Blood pulse | 1 year
  The following vital signs will be recorded according to usual care of COPD and Asthma patient: Pulse (recorded in beat per minute)
Blood pressure | 1 year
  The following vital signs will be recorded according to usual care of COPD and Asthma patient: blood pressure (reported in mmHg)
body temperature | 1 year
  The following vital signs will be recorded according to usual care of COPD and Asthma patient: Body temperature (reported in °C)
respiratory rate | 1 year
  The following vital signs will be recorded according to usual care of COPD and Asthma patient: Respiratory Rate (reported in breath per minute)
St. George Respiratory Questionnaire | 1 year
  Quality of life questionnaires will be collected, according to usual care of COPD and asthma patients.
Asthma control test (ACT) | 1 year
  Quality of life questionnaires will be collected, according to usual care of COPD and asthma patients.
COPD assessment test (CAT) | 1 year
  Quality of life questionnaires will be collected, according to usual care of COPD and asthma patients.

SECONDARY OUTCOMES:
Collection of biological samples | 1 year
  The subject's consent to participate in the genetic research components of the study is not mandatory. Two sputum samples, a total of 20 cc of Bronchoalveolar Lavage (BAL), one sample of bronchoaspirate, one slice of lung biopsies, a total of 15 cc of blood, one sample of stool and a total of 15 cc of urine may be collected during routine clinical practice (at the enrolment visit) on stable state. If for any reason the sample will not be drawn at the inclusion visit, it may be taken at any visit until the last study visit. Samples' collection will be performed once per subject during the study and stored locally at each study site and then sent to the Biobank of the Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico in Milan for storage or to the respiratory Infections Laboratory of the analysis Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico in Milan for analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Blasi, Prof., Principal Investigator — Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico
Locations (4):
- Italy (4):
  - Fondazione IRCCS Cà Granda Ospedale Maggiore Policlinico, Milan, MI
  - Ospedale Papa Giovanni XXIII, Bergamo
  - Ospedale Luigi Sacco, Milano, Milan
  - Fondazione Policlinico Universitario Agostino Gemelli, Roma

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] GBD 2015 Chronic Respiratory Disease Collaborators. Global, regional, and national deaths, prevalence, disability-adjusted life years, and years lived with disability for chronic obstructive pulmonary disease and asthma, 1990-2015: a systematic analysis for the Global Burden of Disease Study 2015. Lancet Respir Med. 2017 Sep;5(9):691-706. doi: 10.1016/S2213-2600(17)30293-X. Epub 2017 Aug 16. PMID 28822787
- [Background] Eapen MS, McAlinden K, Tan D, Weston S, Ward C, Muller HK, Walters EH, Sohal SS. Profiling cellular and inflammatory changes in the airway wall of mild to moderate COPD. Respirology. 2017 Aug;22(6):1125-1132. doi: 10.1111/resp.13021. Epub 2017 Mar 22. PMID 28326668
- [Background] Leung JM, Tiew PY, Mac Aogain M, Budden KF, Yong VF, Thomas SS, Pethe K, Hansbro PM, Chotirmall SH. The role of acute and chronic respiratory colonization and infections in the pathogenesis of COPD. Respirology. 2017 May;22(4):634-650. doi: 10.1111/resp.13032. Epub 2017 Mar 25. PMID 28342288